CLINICAL TRIAL: NCT05741372
Title: Transporter Profiling Study for P-glycoprotein 1 (P-gp), Organic Anion Transporter 1 (OAT1), Organic Anion Transporter 3 (OAT3), Organic Cation Transporter 2 (OCT2), Multidrug and Toxin Extrusion Protein 1 (MATE1), Multidrug and Toxin Extrusion Protein 2-K (MATE2-K), Organic Anion Transporting Polypeptide 1B1 (OATP1B1), Organic Anion Transporting Polypeptide 1B3 (OATP1B3) and Breast Cancer Resistance Protein (BCRP) in Healthy Subjects and in Patients With Stage 4 (F4) Liver Fibrosis / Cirrhosis.
Brief Title: A Study to Compare How Different Medicines (Rosuvastatin, Digoxin, Metformin, and Furosemide) Are Handled by the Body of Healthy People and People With Liver Cirrhosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 0352-2189; 2024-514621-29-00 (Registry Identifier: CTIS)
Record Dates: First submitted 2023-02-14; First posted 2023-02-23 (Actual); Results first posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis | interventions — Rosuvastatin Calcium; Digoxin; Furosemide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1: Healthy participants (Experimental): Healthy participants received a single dose of the following cocktail on Day 1 after a standardized light breakfast and 280 ml of water: 0.25 milligrams (mg) digoxin as tablet, 1 mg furosemide as 0.1 milliliters (ml) oral solution, 10 mg metformin hydrochloride as 0.05 ml oral solution and 10 mg rosuvastatin as film-coated tablet.
  Interventions: Drug: Rosuvastatin; Drug: Digoxin; Drug: Metformin hydrochlorid; Drug: Furosemide
- Group 2: F4 Child-Turcotte-Pugh class A (Child-Pugh A) subjects (compensated) (Experimental): Patients with compensated liver cirrhosis due to any underlying liver disease with advanced fibrosis (F4) and hepatic impairment that meets the criteria for Child-Pugh A received a single dose of the following cocktail on Day 1 after a standardized light breakfast and with 280 ml of water: 0.25 milligrams (mg) digoxin as tablet, 1 mg furosemide as 0.1 milliliters (ml) oral solution, 10 mg metformin hydrochloride as 0.05 ml oral solution and 10 mg rosuvastatin as film-coated tablet.
  Compensated=without any disease symptoms
  Interventions: Drug: Rosuvastatin; Drug: Digoxin; Drug: Metformin hydrochlorid; Drug: Furosemide
- Group 3: F4 Child-Turcotte-Pugh class B (Child-Pugh B) subjects (decompensated) (Experimental): Patients with decompensated liver cirrhosis due to any underlying liver disease with advanced fibrosis (F4) and hepatic impairment that met the criteria for Child-Pugh B received a single dose of the following cocktail on Day 1 after a standardized light breakfast and with 280 ml of water: 0.25 milligrams (mg) digoxin as tablet, 1 mg furosemide as 0.1 milliliters (ml) oral solution, 10 mg metformin hydrochloride as 0.05 ml oral solution and 10 mg rosuvastatin as film-coated tablet.
  Decompensated= with disease symptoms like aszites, variceal bleeding, hepatic encephalopathy, hepato-renal syndrome
  Interventions: Drug: Rosuvastatin; Drug: Digoxin; Drug: Metformin hydrochlorid; Drug: Furosemide

INTERVENTIONS:
Drug: Rosuvastatin — Rosuvastatin
Drug: Digoxin — Digoxin
Drug: Metformin hydrochlorid — Metformin hydrochloride
Drug: Furosemide — Furosemide

SUMMARY:
This study is open to healthy adults and adults with liver cirrhosis. The purpose of this study is to compare how different medicines are handled by the body in people with and without liver cirrhosis. The study measures if the approved medicines rosuvastatin, digoxin, metformin, and furosemide are processed differently in people with liver cirrhosis than in people without liver cirrhosis.

This study will help to understand how new medicines being developed are handled by the body in people with liver cirrhosis. There are 3 groups in this study: people without liver cirrhosis, people with mild liver cirrhosis, and people with moderate liver cirrhosis. All participants get 1 dose each of rosuvastatin, digoxin, metformin, and furosemide by mouth. The participants with liver cirrhosis continue their regular treatment for the condition during the study.

Participants are in the study for about 1 month. During this time, they visit the study site 4 times. For 1 of the visits, they stay overnight for 2 nights at the study site. To assess the main study endpoint, the doctors take frequent blood samples from the participants. The doctors also regularly check participants' health and take note of any unwanted effects.

ELIGIBILITY:
Inclusion criteria

Healthy subjects and F4 liver cirrhosis patients:

* Signed and dated written informed consent in accordance with the International Conference on Harmonization-Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial
* Either male subject, or female subject who meets any of the following criteria for a highly effective contraception from at least 30 days before the first administration of trial medication until 30 days after trial completion:

  * Use of combined (estrogen and progestogen containing) hormonal contraception that prevents ovulation (oral, intravaginal, or transdermal), plus condom
  * Use of progestogen-only hormonal contraception that inhibits ovulation (only injectables or implants), plus condom
  * Use of intrauterine device (IUD) or intrauterine hormone-releasing system (IUS)
  * Sexually abstinent
  * A vasectomized sexual partner who received medical assessment of the surgical success (documented absence of sperm) and provided that the partner is the sole sexual partner of the trial participant
  * Surgically sterilized (including hysterectomy)
  * Postmenopausal, defined as no menses for 1 year without an alternative medical cause (in questionable cases a blood sample with levels of follicle-stimulating hormone (FSH) above 40 units per liter (U/L) and estradiol below 30 nanograms per liter (ng/L) is confirmatory)
  * Not taking any components in the cocktail within 4 weeks of enrolment

Healthy subjects only:

* Healthy male or female subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 75 years (inclusive)
* Body mass index (BMI) of 18.5 to 35 kilograms per meter squared (kg/m2) (inclusive). A BMI of ≥ 30 is no exclusion criterion when the subject can be considered healthy apart from the elevated BMI
* further inclusion criteria apply

F4 liver cirrhosis patients only:

* Male and female subjects, 18 to 75 years
* BMI of 18.5 to 40.0 kg/m2 (inclusive)
* Stable treatment for at least 4 weeks prior to taking the cocktail
* further inclusion criteria apply

Healthy subjects and F4 liver cirrhosis patients:

* Subjects already taking digoxin, furosemide, metformin or rosuvastatin within 4 weeks of enrolment into the study. Furthermore, patients taking ezetimibe, fibrates, or the maximal dose (per Summary of Product Characteristics (SmPC)) of any statin are excluded from this study.
* Subjects with any other condition that would preclude administration of digoxin, furosemide, metformin or rosuvastatin (i.e., contraindicated as per SmPC), such as hypersensitivity to active ingredient or any of the excipients or to sulphonamides, hypovolemia or dehydration, and partial obstructions of urinary outflow (e.g., prostatic hypertrophy)
* Repeated measurement of systolic blood pressure outside the range of 90 to 150 millimeter of mercury (mmHg), diastolic blood pressure outside the range of 50 to 95 mmHg, or pulse rate outside the range of 60 to 90 beats per minute (bpm)
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Relevant (other than Hepatitis B virus (HBV) or Hepatitis C virus (HCV)) chronic or acute infections (including an ongoing severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection)
* Patients receiving antiviral therapy at the time of inclusion into the trial
* further exclusion criteria apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2023-09-07 (Actual); Primary Completion 2024-12-18 (Actual); Study Completion 2024-12-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- CRS Clinical Research Services Mannheim GmbH, Mannheim, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g., studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization). For more details refer to: https:// www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The purpose of this single dose, open label study was to investigate whether the maximum concentration (Cmax) and the area under the concentration-time curve of the analyte in plasma from time point 0 to time point 24 hours (AUC0-24) values for the different components in the transporter cocktail - digoxin, furosemide, metformin and rosuvastatin are similar or different in F4 graded liver fibrosis (cirrhosis) patients on standard therapy compared to healthy participants.
Pre-assignment Details: Only subjects that met all the study inclusion and none of the exclusion criteria were to be entered in the study. All subjects were free to withdraw from the clinical trial at any time for any reason given. Close monitoring of all subjects was adhered to throughout the trial conduct. Rescue medication was allowed for all patients as required.
Period: Overall Study
Arm/Group | Group 1: Healthy Participants | Group 2: F4 Child-Turcotte-Pugh Class A (Child-Pugh A) Subjects (Compensated) | Group 3: F4 Child-Turcotte-Pugh Class B (Child-Pugh B) Subjects (Decompensated)
Started | 11 | 11 | 6
Completed | 11 | 11 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): The treated set included all subjects who signed informed consent and were treated with at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Healthy Participants | Group 2: F4 Child-Turcotte-Pugh Class A (Child-Pugh A) Subjects (Compensated) | Group 3: F4 Child-Turcotte-Pugh Class B (Child-Pugh B) Subjects (Decompensated) | Total
Number analyzed (Participants) | 11 | 11 | 6 | 28
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.5 (8.9) | 60.2 (11.9) | 61.2 (13.5) | 59.7 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 2 | 14
  Male | 5 | 5 | 4 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 11 | 11 | 6 | 28
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 11 | 11 | 6 | 28
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration Time Curve of Rosuvastatin in Plasma Over the Time Interval From 0 to 24 Hours (AUC0-24)
Description: Adjusted geometric means and adjusted geometric standard errors were calculated using an analysis of variance (ANOVA) model on the logarithmic scale.
  The pharmacokinetics endpoint was log transformed (natural logarithm) prior to fitting the ANOVA model. This model included effects accounting for the following sources of variation: 'group', age, and BMI. All effects were considered as fixed.
Time Frame: Within 2 hours (hrs) before and at 30 minutes (min), 1 hrs, 1.5 hrs, 2 hrs, 3 hrs, 4 hrs, 6 hrs, 8 hrs, 10 hrs, 12 hrs, and 24 hrs after drug administration.
Population: Pharmacokinetic parameter analysis set (PKS): This set included all subjects in the treated set (TS) who provided at least one pharmacokinetics (PK) endpoint that was defined as primary and was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability. Descriptive and model-based analyses of PK parameters were based on the PKS.
Measure: Geometric Least Squares Mean (Standard Error); unit: hours*nanomole/liters (h*nmol/l)
Arm/Group | Group 1: Healthy Participants | Group 2: F4 Child-Turcotte-Pugh Class A (Child-Pugh A) Subjects (Compensated) | Group 3: F4 Child-Turcotte-Pugh Class B (Child-Pugh B) Subjects (Decompensated)
Number analyzed (Participants) | 11 | 11 | 6
hours*nanomole/liters (h*nmol/l) | 94.5 (NA) — NA = adjusted geometric standard error = 1.18 | 120.2 (NA) — NA = adjusted geometric standard error = 1.18 | 704.6 (NA) — NA = adjusted geometric standard error = 1.25
Statistical Analysis 1: Comparison: Group 1: Healthy Participants vs Group 2: F4 Child-Turcotte-Pugh Class A (Child-Pugh A) Subjects (Compensated); The adjusted geometric means ratio based on ANOVA was calculated by using least square means, the 90% CI by using residual error from quantiles from t-distribution. These quantities were back-transformed to original scale; Test type: Other; Adjusted geometric mean ratio = 127.2, 90% CI 2-sided [85.4 to 189.6] — Ratio [%]=(adjusted geometric mean Group 2/adjusted geometric mean Group 1)*100. Total gCV = 23.6%
Statistical Analysis 2: Comparison: Group 1: Healthy Participants vs Group 3: F4 Child-Turcotte-Pugh Class B (Child-Pugh B) Subjects (Decompensated); [analysis description as in outcome 1, analysis 1]; Test type: Other; Adjusted geometric mean ratio = 745.7, 90% CI 2-sided [464.9 to 1196] — Ratio [%]=(adjusted geometric mean Group 3/adjusted geometric mean Group 1)*100. Total gCV = 28.1%

2. Primary Outcome: Maximum Measured Concentration of Rosuvastatin in Plasma (Cmax)
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Standard Error); unit: nanomole/liters (nmol/l)
Groups:
- Group 1: Healthy Participants: Healthy participants received a single dose of the following cocktail on Day 1 after a standardized light breakfast and 280 ml of water: O.25 milligrams (mg) digoxin as tablet, 1 mg furosemide as 0.1 milliliters (ml) oral solution, 10 mg metformin hydrochloride as 0.05 ml oral solution and 10 mg rosuvastatin as film-coated tablet.
- Group 2: F4 Child-Turcotte-Pugh Class A (Child-Pugh A) Subjects (Compensated): Patients with compensated liver cirrhosis due to any underlying liver disease with advanced fibrosis (F4) and hepatic impairment that meets the criteria for Child-Pugh A received a single dose of the following cocktail on Day 1 after a standardized light breakfast and with 280 ml of water: O.25 milligrams (mg) digoxin as tablet, 1 mg furosemide as 0.1 milliliters (ml) oral solution, 10 mg metformin hydrochloride as 0.05 ml oral solution and 10 mg rosuvastatin as film-coated tablet.
  Compensated=without any disease symptoms
- Group 3: F4 Child-Turcotte-Pugh Class B (Child-Pugh B) Subjects (Decompensated): Patients with decompensated liver cirrhosis due to any underlying liver disease with advanced fibrosis (F4) and hepatic impairment that met the criteria for Child-Pugh B received a single dose of the following cocktail on Day 1 after a standardized light breakfast and with 280 ml of water: O.25 milligrams (mg) digoxin as tablet, 1 mg furosemide as 0.1 milliliters (ml) oral solution, 10 mg metformin hydrochloride as 0.05 ml oral solution and 10 mg rosuvastatin as film-coated tablet.
  Decompensated= with disease symptoms like aszites, variceal bleeding, hepatic encephalopathy, hepato-renal syndrome
Arm/Group | Group 1: Healthy Participants | Group 2: F4 Child-Turcotte-Pugh Class A (Child-Pugh A) Subjects (Compensated) | Group 3: F4 Child-Turcotte-Pugh Class B (Child-Pugh B) Subjects (Decompensated)
Number analyzed (Participants) | 11 | 11 | 6
nanomole/liters (nmol/l) | 9.8 (NA) — NA = adjusted geometric standard error = 1.20 | 17.9 (NA) — NA = adjusted geometric standard error = 1.20 | 167.1 (NA) — NA = adjusted geometric standard error = 1.28
Statistical Analysis 1: Comparison: Group 1: Healthy Participants vs Group 2: F4 Child-Turcotte-Pugh Class A (Child-Pugh A) Subjects (Compensated); [analysis description as in outcome 1, analysis 1]; Test type: Other; Adjusted geometric mean ratio = 183.6, 90% CI 2-sided [117.3 to 287.5] — Ratio [%]=(adjusted geometric mean Group 2/adjusted geometric mean Group 1)*100. Total gCV = 26.6%
Statistical Analysis 2: Comparison: Group 1: Healthy Participants vs Group 3: F4 Child-Turcotte-Pugh Class B (Child-Pugh B) Subjects (Decompensated); [analysis description as in outcome 1, analysis 1]; Test type: Other; Adjusted geometric mean ratio = 1712.2, 90% CI 2-sided [1006.7 to 2912.2] — Ratio [%]=(adjusted geometric mean Group 3/adjusted geometric mean Group 1)*100. Total gCV = 31.7%

3. Primary Outcome: Area Under the Concentration Time Curve of Digoxin in Plasma Over the Time Interval From 0 to 24 Hours (AUC0-24)
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Standard Error); unit: hours*nanomole/liters (h*nmol/l)
Arm/Group | Group 1: Healthy Participants | Group 2: F4 Child-Turcotte-Pugh Class A (Child-Pugh A) Subjects (Compensated) | Group 3: F4 Child-Turcotte-Pugh Class B (Child-Pugh B) Subjects (Decompensated)
Number analyzed (Participants) | 11 | 11 | 6
hours*nanomole/liters (h*nmol/l) | 8.1 (NA) — NA = adjusted geometric standard error = 1.08 | 7.8 (NA) — NA = adjusted geometric standard error = 1.08 | 7.6 (NA) — NA = adjusted geometric standard error = 1.10
Statistical Analysis 1: Comparison: Group 1: Healthy Participants vs Group 2: F4 Child-Turcotte-Pugh Class A (Child-Pugh A) Subjects (Compensated); [analysis description as in outcome 1, analysis 1]; Test type: Other; Adjusted geometric mean ratio = 96.6, 90% CI 2-sided [81.0 to 115.3] — Ratio [%]=(adjusted geometric mean Group 2/adjusted geometric mean Group 1)*100. Total gCV = 10.3%
Statistical Analysis 2: Comparison: Group 1: Healthy Participants vs Group 3: F4 Child-Turcotte-Pugh Class B (Child-Pugh B) Subjects (Decompensated); [analysis description as in outcome 1, analysis 1]; Test type: Other; Adjusted geometric mean ratio = 93.6, 90% CI 2-sided [75.9 to 115.3] — Ratio [%]=(adjusted geometric mean Group 3/adjusted geometric mean Group 1)*100. Total gCV = 12.2%

4. Primary Outcome: Maximum Measured Concentration of Digoxin in Plasma (Cmax)
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Standard Error); unit: nanomole/liters (nmol/l)
Arm/Group | Group 1: Healthy Participants | Group 2: F4 Child-Turcotte-Pugh Class A (Child-Pugh A) Subjects (Compensated) | Group 3: F4 Child-Turcotte-Pugh Class B (Child-Pugh B) Subjects (Decompensated)
Number analyzed (Participants) | 11 | 11 | 6
nanomole/liters (nmol/l) | 1.7 (NA) — NA = adjusted geometric standard error = 1.09 | 1.3 (NA) — NA = adjusted geometric standard error = 1.09 | 1.4 (NA) — NA = adjusted geometric standard error = 1.13
Statistical Analysis 1: Comparison: Group 1: Healthy Participants vs Group 2: F4 Child-Turcotte-Pugh Class A (Child-Pugh A) Subjects (Compensated); [analysis description as in outcome 1, analysis 1]; Test type: Other; Adjusted geometric mean ratio = 78.9, 90% CI 2-sided [63.8 to 97.5] — Ratio [%]=(adjusted geometric mean Group 2/adjusted geometric mean Group 1)*100. Total gCV = 12.5%
Statistical Analysis 2: Comparison: Group 1: Healthy Participants vs Group 3: F4 Child-Turcotte-Pugh Class B (Child-Pugh B) Subjects (Decompensated); [analysis description as in outcome 1, analysis 1]; Test type: Other; Adjusted geometric mean ratio = 83.6, 90% CI 2-sided [65.0 to 107.5] — Ratio [%]=(adjusted geometric mean Group 3/adjusted geometric mean Group 1)*100. Total gCV = 14.8%

5. Primary Outcome: Area Under the Concentration Time Curve of Metformin in Plasma Over the Time Interval From 0 to 24 Hours (AUC0-24)
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Standard Error); unit: hours*nanomole/liters (h*nmol/l)
Arm/Group | Group 1: Healthy Participants | Group 2: F4 Child-Turcotte-Pugh Class A (Child-Pugh A) Subjects (Compensated) | Group 3: F4 Child-Turcotte-Pugh Class B (Child-Pugh B) Subjects (Decompensated)
Number analyzed (Participants) | 11 | 11 | 6
hours*nanomole/liters (h*nmol/l) | 2035.7 (NA) — NA = adjusted geometric standard error = 1.07 | 1982.8 (NA) — NA = adjusted geometric standard error = 1.07 | 1917.9 (NA) — NA = adjusted geometric standard error = 1.09
Statistical Analysis 1: Comparison: Group 1: Healthy Participants vs Group 2: F4 Child-Turcotte-Pugh Class A (Child-Pugh A) Subjects (Compensated); [analysis description as in outcome 1, analysis 1]; Test type: Other; Adjusted geometric mean ratio = 97.4, 90% CI 2-sided [83.2 to 114] — Ratio [%]=(adjusted geometric mean Group 2/adjusted geometric mean Group 1)*100. Total gCV = 9.2%
Statistical Analysis 2: Comparison: Group 1: Healthy Participants vs Group 3: F4 Child-Turcotte-Pugh Class B (Child-Pugh B) Subjects (Decompensated); [analysis description as in outcome 1, analysis 1]; Test type: Other; Adjusted geometric mean ratio = 94.2, 90% CI 2-sided [78.2 to 113.5] — Ratio [%]=(adjusted geometric mean Group 3/adjusted geometric mean Group 1)*100. Total gCV = 10.9%

6. Primary Outcome: Maximum Measured Concentration of Metformin in Plasma (Cmax)
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Standard Error); unit: nanomole/liters (nmol/l)
Arm/Group | Group 1: Healthy Participants | Group 2: F4 Child-Turcotte-Pugh Class A (Child-Pugh A) Subjects (Compensated) | Group 3: F4 Child-Turcotte-Pugh Class B (Child-Pugh B) Subjects (Decompensated)
Number analyzed (Participants) | 11 | 11 | 6
nanomole/liters (nmol/l) | 348.0 (NA) — NA = adjusted geometric standard error = 1.07 | 303.6 (NA) — NA = adjusted geometric standard error = 1.07 | 291.0 (NA) — NA = adjusted geometric standard error = 1.10
Statistical Analysis 1: Comparison: Group 1: Healthy Participants vs Group 2: F4 Child-Turcotte-Pugh Class A (Child-Pugh A) Subjects (Compensated); [analysis description as in outcome 1, analysis 1]; Test type: Other; Adjusted geometric mean ratio = 87.3, 90% CI 2-sided [74.0 to 102.9] — Ratio [%]=(adjusted geometric mean Group 2/adjusted geometric mean Group 1)*100. Total gCV = 9.7%
Statistical Analysis 2: Comparison: Group 1: Healthy Participants vs Group 3: F4 Child-Turcotte-Pugh Class B (Child-Pugh B) Subjects (Decompensated); [analysis description as in outcome 1, analysis 1]; Test type: Other; Adjusted geometric mean ratio = 83.6, 90% CI 2-sided [68.8 to 101.7] — Ratio [%]=(adjusted geometric mean Group 3/adjusted geometric mean Group 1)*100. Total gCV = 11.5%

7. Primary Outcome: Area Under the Concentration Time Curve of Furosemide in Plasma Over the Time Interval From 0 to 24 Hours (AUC0-24)
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Standard Error); unit: hours*nanomole/liters (h*nmol/l)
Arm/Group | Group 1: Healthy Participants | Group 2: F4 Child-Turcotte-Pugh Class A (Child-Pugh A) Subjects (Compensated) | Group 3: F4 Child-Turcotte-Pugh Class B (Child-Pugh B) Subjects (Decompensated)
Number analyzed (Participants) | 11 | 11 | 6
hours*nanomole/liters (h*nmol/l) | 238.0 (NA) — NA = adjusted geometric standard error = 1.09 | 210.1 (NA) — NA = adjusted geometric standard error = 1.09 | 275.0 (NA) — NA = adjusted geometric standard error = 1.12
Statistical Analysis 1: Comparison: Group 1: Healthy Participants vs Group 2: F4 Child-Turcotte-Pugh Class A (Child-Pugh A) Subjects (Compensated); [analysis description as in outcome 1, analysis 1]; Test type: Other; Adjusted geometric mean ratio = 88.3, 90% CI 2-sided [71.6 to 108.8] — Ratio [%]=(adjusted geometric mean Group 2/adjusted geometric mean Group 1)*100. Total gCV = 12.2%
Statistical Analysis 2: Comparison: Group 1: Healthy Participants vs Group 3: F4 Child-Turcotte-Pugh Class B (Child-Pugh B) Subjects (Decompensated); [analysis description as in outcome 1, analysis 1]; Test type: Other; Adjusted geometric mean ratio = 115.5, 90% CI 2-sided [90.2 to 148.0] — Ratio [%]=(adjusted geometric mean Group 3/adjusted geometric mean Group 1)*100. Total gCV = 14.5%

8. Primary Outcome: Maximum Measured Concentration of Furosemide in Plasma (Cmax)
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Standard Error); unit: nanomole/liters (nmol/l)
Arm/Group | Group 1: Healthy Participants | Group 2: F4 Child-Turcotte-Pugh Class A (Child-Pugh A) Subjects (Compensated) | Group 3: F4 Child-Turcotte-Pugh Class B (Child-Pugh B) Subjects (Decompensated)
Number analyzed (Participants) | 11 | 11 | 6
nanomole/liters (nmol/l) | 81.1 (NA) — NA = adjusted geometric standard error = 1.10 | 62.3 (NA) — NA = adjusted geometric standard error = 1.10 | 78.0 (NA) — NA = adjusted geometric standard error = 1.14
Statistical Analysis 1: Comparison: Group 1: Healthy Participants vs Group 2: F4 Child-Turcotte-Pugh Class A (Child-Pugh A) Subjects (Compensated); [analysis description as in outcome 1, analysis 1]; Test type: Other; Adjusted geometric mean ratio = 76.8, 90% CI 2-sided [61.1 to 96.6] — Ratio [%]=(adjusted geometric mean Group 2/adjusted geometric mean Group 1)*100. Total gCV = 13.4%
Statistical Analysis 2: Comparison: Group 1: Healthy Participants vs Group 3: F4 Child-Turcotte-Pugh Class B (Child-Pugh B) Subjects (Decompensated); [analysis description as in outcome 1, analysis 1]; Test type: Other; Adjusted geometric mean ratio = 96.2, 90% CI 2-sided [73.4 to 126.1] — Ratio [%]=(adjusted geometric mean Group 3/adjusted geometric mean Group 1)*100. Total gCV = 15.9%

ADVERSE EVENTS:
Time Frame: For AEs on-treatment period: From start of drug administration on Day 1 plus longest residual effect period for drugs in the cocktail, up to 10 days. For all-cause mortality: From start of drug administration until end of follow-up, up to 18 days.
Description: Treated set (TS): The treated set included all subjects who signed informed consent and were treated with at least one dose of study drug. The treated set was used for safety analyses.
Arm/Group | Group 1: Healthy Participants | Group 2: F4 Child-Turcotte-Pugh Class A (Child-Pugh A) Subjects (Compensated) | Group 3: F4 Child-Turcotte-Pugh Class B (Child-Pugh B) Subjects (Decompensated)
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11 | 0/6
Other Adverse Events (participants affected / at risk) | 3/11 | 3/11 | 0/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: Healthy Participants (N=11) | Group 2: F4 Child-Turcotte-Pugh Class A (Child-Pugh A) Subjects (Compensated) (N=11) | Group 3: F4 Child-Turcotte-Pugh Class B (Child-Pugh B) Subjects (Decompensated) (N=6)
Headache (Nervous system disorders) | 2 | 2 | 0
Taste disorder (Nervous system disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2023-03-09): https://cdn.clinicaltrials.gov/large-docs/72/NCT05741372/Prot_000.pdf
  • Statistical Analysis Plan (2025-03-17): https://cdn.clinicaltrials.gov/large-docs/72/NCT05741372/SAP_001.pdf